CLINICAL TRIAL: NCT00574262
Title: Quality of Acute Stroke Care Evaluated With a Clinical Pathway on a 16 Bed Stroke Unit - a Prospective Trial
Brief Title: Quality Assessment in Acute Stroke Care
Acronym: QuASt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Prof. Dr. Wolf-Rüdiger Schäbitz, Department of Neurology, University Hospital Muenster
Other Study IDs: ClinPathStroke
Record Dates: First submitted 2007-11-23; First posted 2007-12-17 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2007-11

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; clinical pathway; quality of care; secondary prevention
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to evaluate the quality of care on a 16 bed stroke unit by using a new developed clinical pathway.

ELIGIBILITY:
Inclusion Criteria:

* admission to the stroke unit of the university hospital in Muenster, Germany
* acute ischemic stroke or transient ischemic attack

Exclusion Criteria:

* intracerebral haemorrhage
* neurological symptoms due to other pathology than acute ischemic stroke or transient ischemic attack
* intraarterial thrombolysis
* necessity of artificial ventilation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with an acute ischemic stroke admitted to the stroke unit of the university hospital in Muenster, Germany
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-10; Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
frequency of patients monitored according to the specific german procedure standard (OPS-code 8-981) (preset target 90 - 95 %) | duration of stay on stroke unit

SECONDARY OUTCOMES:
frequency of stroke been classified according to the TOAST criteria (preset target 55 - 65 %) | duration of stay on stroke unit
frequency of initiated or improved antithrombotic secondary prevention (preset target 90 - 95 %) | duration of stay on stroke unit
frequency of initiated or improved statin therapy (preset target 40 - 50 %) | duration of stay on stroke unit
frequency of totally completed clinical diagnostics regarding the etiology of the stroke (preset target 60 -70 %) | duration of stay on stroke unit
frequency of initiated or improved antihypertension therapy and reduction of systolic and diastolic blood pressure by more than 10 mmHg (preset target 60 - 70 %) | duration of stay on stroke unit
frequency of a reduction on the NIH-SS by at least two points (preset target 50 - 60 %) | duration of stay on stroke unit

CONTACTS AND LOCATIONS:
Overall Officials: Wolf Rüdiger Schäbitz, MD, Principal Investigator — Department of Neurology, University Hospital of Muenster, Germany
Locations (1):
- Department of Neurology, University Hospital of Muenster, Münster, Germany

REFERENCES:
- [Background] Heuschmann PU, Biegler MK, Busse O, Elsner S, Grau A, Hasenbein U, Hermanek P, Janzen RW, Kolominsky-Rabas PL, Kraywinkel K, Lowitzsch K, Misselwitz B, Nabavi DG, Otten K, Pientka L, von Reutern GM, Ringelstein EB, Sander D, Wagner M, Berger K. Development and implementation of evidence-based indicators for measuring quality of acute stroke care: the Quality Indicator Board of the German Stroke Registers Study Group (ADSR). Stroke. 2006 Oct;37(10):2573-8. doi: 10.1161/01.STR.0000241086.92084.c0. Epub 2006 Sep 7. PMID 16960092
- [Background] Kwan J. Care pathways for acute stroke care and stroke rehabilitation: from theory to evidence. J Clin Neurosci. 2007 Mar;14(3):189-200. doi: 10.1016/j.jocn.2006.01.026. PMID 17258128
- [Background] Taylor WJ, Wong A, Siegert RJ, McNaughton HK. Effectiveness of a clinical pathway for acute stroke care in a district general hospital: an audit. BMC Health Serv Res. 2006 Feb 23;6:16. doi: 10.1186/1472-6963-6-16. PMID 16504101